CLINICAL TRIAL: NCT01098058
Title: A Proof of Concept Randomised Controlled Trial to Examine the Potential Efficacy, Patient Acceptability and Feasibility of Cognitive-behavioural Therapy for Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Cognitive-Behavioural Therapy (CBT) for Adult Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Antonia Dittner, Senior Clinical Psychologist, South London and Maudsley NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/H0721/49
Record Dates: First submitted 2010-03-19; First posted 2010-04-02 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Adult attention deficit hyperactivity disorder; cognitive-behavioural therapy; randomised controlled trial
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT plus treatment as usual (Experimental)
  Interventions: Other: CBT plus treatment as usual
- Treatment as usual (Active Comparator): Treatment as usual appointments at the Adult ADHD Service - typically one 30-minute appointment every three to six months
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: CBT plus treatment as usual — 16 one-hour therapy sessions taking place over 42 weeks in addition to usual medical follow-up appointments
  Arms: CBT plus treatment as usual
Other: Treatment as usual — Treatment as usual appointments at the Adult ADHD Service - typically one 30-minute appointment every three to six months
  Arms: Treatment as usual

SUMMARY:
The purpose of the study is to compare the effectiveness of cognitive-behavioural therapy (CBT) plus treatment as usual with treatment as usual only in treating adults with attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
Approximately 50% of individuals with adult ADHD are not able to tolerate, do not respond to, or fail to reach optimal outcomes on medication alone (Spencer, Biederman and Wilens 2000). The NICE guidelines for adult ADHD, released in September 2008, emphasise the need for further such research into psychological approaches to treatment of the condition.

There is promising preliminary evidence that suggests that psychological approaches to treatment are effective in individuals with Adult ADHD (see Weiss et al 2008 for a review). So far, however, only one randomised controlled trial of CBT has been carried out (Safren, Otto et al 2005). Thirty-one participants were randomised to receive either CBT and medication as usual or medication alone. Those randomised to CBT (n=16) had significantly lower ADHD symptoms (as rated by an independent investigator), global severity and self-rated symptoms than those on medication only (ps range <0.01 to <0.002). Those in the CBT group also had significantly lower scores on independently- and self-rated measures of mood (ps range <0.01 to 0.04).

There is a need for more randomised controlled trials to be carried out in order to replicate Safren et al's result in a different site, to further investigate the feasibility of CBT in this population and to further develop CBT approaches to this condition.

Studies carried out so far have tended to be skills-based (i.e. sessions focused on teaching specific skills such as time management), rather than formulation-driven (a formulation is essentially a shared hypothesis as to the relationships between the individual's experience, beliefs, behaviour and emotions).

The current study aims to evaluate a formulation-driven approach to CBT for adults with ADHD. A group of individuals (n = 30) receiving CBT combined with treatment as usual for adults with ADHD will be compared with a group receiving treatment as usual only (n= 30), employing a randomized design.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of adult ADHD according to NICE guidelines i.e. if there was evidence from both the participant and the informant (where available) that 1) the participant met DSM-IV criteria for Adult ADHD both in childhood and adulthood 2) that they experienced at least moderate psychological, social and/or educational or occupational impairment in multiple settings and 3) symptoms occurred in two or more settings including social, familial, educational and/or occupational settings. Participants will have received a diagnosis either from the Adult ADHD Service, Maudsley Hospital, London, UK or another specialist/secondary care service (in this case a copy of the diagnostic report will be required). Participants will either already be attending follow-up clinics, including psychoeducation workshops, or will have been recently referred to the service for medication follow-up or psychological treatment.
* Currently score 6 or more on the inattentive or hyperactive/impulsive subscale of the Adult Barkley Current Behaviour Scale
* Clinical severity of at least a moderate level (Clinical Global Impression score of 4 or above)
* Able to attend the clinic regularly and reliably

Exclusion Criteria:

* Clinically significant anxiety disorder
* Current episode major depression, current suicidality or self-harm (score of moderate or high suicidality on the M.I.N.I.)
* Acquired brain injury
* Primary diagnosis of psychosis or bipolar disorder
* Pervasive developmental disorder(score of <= 32 on Autism Spectrum Quotient - although if the assessor judges that items that confound with ADHD have caused the score to be elevated, people with scores >=32 can still enter the trial)
* Diagnosis of personality disorder
* Active substance misuse/dependence in last three months
* Verbal IQ <80
* Not able to comply with the requirements of a randomised controlled trial
* If the assessor does not perceive ADHD to be the primary problem

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Adult Barkley Current Behaviour Scale (Barkley 2006) | week 42
  18-item self-report measure assessing ADHD symptoms, rated on a 4-point Likert scale
Work and Social Adjustment Scale (Mundt et al 2002) | week 42
  A reliable and valid self-report measure of impaired functioning attributable to an identified problem.
  It consists of 5 items, each rated on an 8-point scale

SECONDARY OUTCOMES:
Clinical Global Impression Scales (Guy 1976) | week 42
  The Clinical Global Impression Scale is a 7-point scale that requires the clinician to rate the current severity of the patient's illness , relative to the past experience with patients with the same diagnosis. It is widely used in clinical treatment trials and is reliable and valid.
  There are severity, improvement and satisfaction versions of the scale. Clinician, independent evaluator will complete severity measure. Participant, clinician, independent evaluator and informant will complete improvement measure; participant will complete satisfaction measure.
Clinical Outcomes in Routine Evaluation (CORE-OM) (Evans et al 2002) | week 42
  The CORE-OM is a standardised public domain approach to audit, evaluation and outcome measurement for UK psychological therapy and counselling services. It consists of 34 items measured on a five-point Likert scale and assesses emotional distress and risk over the past week.
Hospital anxiety and depression scale (Zigmond and Snaith 1983) | week 42
  A reliable and valid 14-item self-report scale assessing anxiety and depression symptoms, scored on a 4-point likert scale.
ADHD Beliefs Questionnaire | week 42
  The ADHD Beliefs Questionnaire is a measure designed for the study. It consists of 28 items measured on a 5-point Likert Scale. Questions relate to specific beliefs that clinically have been noted to be associated with adult ADHD, e.g. "my lack of concentration will stop me achieving the things that I want".
ADHD Behaviours Questionnaire | week 42
  The ADHD Behaviours Questionnaire is a measure designed for the study. It consists of 29 items measured on a 5-point Likert Scale. Questions relate to specific behaviours that clinically have been noted to be associated with adult ADHD, e.g. "I avoid or put off doing things that I do not find interesting".
Rosenberg Self-Esteem Scale (Rosenberg 1965) | week 42
  The Rosenberg Self-Esteem Scale is a 10-item self-report measure of global self-esteem. It consists of 10 statements related to overall feelings of self-worth or self-acceptance. The items are answered on a four-point scale ranging from strongly agree to strongly disagree.
Informant-rated Adult Barkley Current Behaviour Scale (Barkley 2006) | week 42
  This is the same as the Adult Barkley Current Behaviour scale but adapted to be completed by an informant.
Global assessment of functioning scale, DSM IV-TR | week 42
  The Global Assessment of Functioning (GAF) is a numeric scale (0 through 100) used by mental health clinicians and physicians to subjectively rate the social, occupational, and psychological functioning of adults.
Frost Multidimensional Perfectionism Scale (Frost et al 1990), Doubts about actions, Concern over mistakes, Parental Criticism and Parental expectations subscales | Week 42
  22 items, each measured on a 5-point Likert scale. The scale has good reliability and validity.
Beliefs about Emotions Questionnaire (Rimes et al 2009) | week 42
  The scale has 12 items assessed on a 7-point Likert scale. It has good reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia J Dittner, D Clin Psy, Principal Investigator — South London and Maudsley NHS Foundation Trust
Locations (1):
- Adult ADHD Service, South London and Maudsley NHS Foundation Trust, London, London, United Kingdom

REFERENCES:
- [Background] Barkley R.A. (2006) Attention-Deficit Hyperactivity Disorder - A Handbook for Diagnosis and Treatment. Third Edition, The Guildford Press, New York.
- [Background] Rosenberg, M. (1965). Society and The Adolescent Self-Image. Princeton, N.J.: Princeton University Press.
- [Background] Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR). American Psychiatric Association, 2000.
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Evans C, Connell J, Barkham M, Margison F, McGrath G, Mellor-Clark J, Audin K. Towards a standardised brief outcome measure: psychometric properties and utility of the CORE-OM. Br J Psychiatry. 2002 Jan;180:51-60. doi: 10.1192/bjp.180.1.51. PMID 11772852
- [Background] Guy W (ed). ECDEU Assessment Manual for Psychopharmacology. Rockville, MD: US Department of Heath, Education, and Welfare Public Health Service Alcohol, Drug Abuse, and Mental Health Administration, 1976.
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645